CLINICAL TRIAL: NCT04128280
Title: Multi-center Clinical Observation of a New Treatment Method Based on the Pathogenesis of Obstructive Prostatitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Sir Run Run Shaw Hospital (Other); Xin Hua Hospital of Zhejiang Province (Other); Huashan Hospital (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Changhai Hospital (Other); Peking University First Hospital (Other); The First Affiliated Hospital of Shanxi Medical University (Other); The Affiliated Hospital of Qingdao University (Other); First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-307
Record Dates: First submitted 2019-10-14; First posted 2019-10-16 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2019-10

CONDITIONS: Chronic Prostatitis
Keywords: Chronic Prostatitis
MeSH Terms: interventions — tubercidin-5'-diphosphate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (Experimental): Test group: Patients will receive a surgery: transurethral dilation of prostate with a columnar balloon
  Interventions: Procedure: TUDP
- Control Group (Active Comparator): Control group: Patients will receive a surgery: transurethral incision of bladder neck.
  Interventions: Procedure: TUIB

INTERVENTIONS:
Procedure: TUDP — a surgery: transurethral dilation of prostate with a columnar balloon
  Arms: Test Group
Procedure: TUIB — a surgery: transurethral incision of bladder neck
  Arms: Control Group

SUMMARY:
Multi-center clinical observation of a new treatment method based on the pathogenesis of obstructive prostatitis

DETAILED DESCRIPTION:
1. Study purpose: To investigate the therapeutic effect of transurethral dilation of prostate with a columnar balloon on patients with chronic obstructive prostatitis
2. Study design: A randomized, controlled, multi-center clinical trial
3. Study subjects: Patients with chronic obstructive prostatitis
4. Number of subjects: 180
5. Surgery treatments:

Test group: Patients will receive a surgery: transurethral dilation of prostate with a columnar balloon.

Control group: Patients will receive a surgery: transurethral incision of bladder neck.

ELIGIBILITY:
Inclusion Criteria:

1. older than 35 years old, urinary obstruction is clear;
2. the total score of chronic prostatitis symptoms index (CPSI) is greater than 14 points, and the severity of symptoms is greater than 9 points;
3. maximum urine flow rate is less than 15 ml/s;
4. cystoscopy and pathological biopsy confirmed the presence of bladder neck fibrosis, bladder trabeculae formation;
5. other conservative treatments are ineffective or ineffective, and drug treatment is not effective for more than 6 months;
6. voluntarily participated in this clinical trial, complied with the requirements of this study and signed the informed consent form.

Exclusion Criteria:

1. urinary tract infection, urinary tumor, history of intestinal inflammatory disease;
2. neurogenic bladder;
3. history of pelvic radiation therapy or chemotherapy;
4. PSA is abnormal;
5. urethral stricture, history of bladder or prostate surgery;
6. the investigator determined that it is not suitable for this clinical trial.

Ages: 35 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
The score of CPSI | within 12 months after surgery
  measure the chronic prostatitis symptom index (CPSI) by a questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China